CLINICAL TRIAL: NCT07199738
Title: A Multi-Center Study Assessing the Safety and Efficacy of the LEGION Medial Stabilized (MS) Insert in Patients Undergoing a Total Knee Arthroplasty (TKA)
Status: Not yet recruiting | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SNIS-O-1285
Record Dates: First submitted 2025-08-28; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-07

CONDITIONS: Inflammatory Arthritis; Primary Total Knee Arthroplasty Due to Degenerative Joint Disease (Primary Diagnosis of Osteoarthritis); Post-traumatic Arthritis
Keywords: Primary TKA; Osteoarthritis; post-traumatic arthritis; inflammatory arthritis
MeSH Terms: conditions — Arthritis; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Cemented CoCr: LEGION MS with Cemented Tibia (JII) with LEGION CR non-porous (CoCr) Femoral component
  Interventions: Device: Cemented CoCr
- Cemented Oxinium: LEGION MS with Cemented Tibia (JII) with LEGION CR non-porous (Ox) Femoral component
  Interventions: Device: Cemented Oxinium
- Cementless: LEGION MS with CONCELOC Tibia with LEGION CR porous (without HA) Femoral component
  Interventions: Device: Cementless

INTERVENTIONS:
Device: Cemented CoCr — Primary TKA performed using the LEGION MS with Cemented Tibia (JII) with LEGION CR non-porous (CoCr) Femoral component
  Groups: Cemented CoCr
Device: Cemented Oxinium — Primary TKA performed using the LEGION MS with Cemented Tibia (JII) with LEGION CR non-porous (Ox) Femoral component
  Groups: Cemented Oxinium
Device: Cementless — Primary TKA performed using the LEGION MS with CONCELOC Tibia with LEGION CR porous (without HA) Femoral component
  Groups: Cementless

SUMMARY:
The purpose of this study is to assess the long-term safety and performance of the LEGION Medial Stabilized insert and to generate clinical evidence to support and maintain product registration in global markets.

DETAILED DESCRIPTION:
This is a post market, prospective and retro-prospective, multicentered 10-year observational study. The study is looking at the LEGION Medial Stabilized insert used in primary total knee arthroplasty alongside specific tibia and femur component combinations. There will be 144 knees enrolled across 3 cohorts in the study. All enrolled knees will undergo a primary knee arthroplasty due to degenerative joint disease (primary diagnosis of osteoarthritis), post-traumatic arthritis or inflammatory arthritis. Enrolled subjects will be followed up for 10 years post operation.

ELIGIBILITY:
Inclusion Criteria:

1. A). Prospective Subjects: Subject needing primary Total Knee Arthroplasty (TKA) due to degenerative joint disease (primary diagnosis of osteoarthritis), post-traumatic arthritis or inflammatory arthritis.

   OR

   B). Retro-prospective Subjects: Subject has undergone primary TKA using the investigational product in the past 12 months to repair degenerative joint disease, post-traumatic arthritis or inflammatory arthritis and all the following conditions have been met:
   * Pre-operative Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS JR) has been obtained
   * Post-operative radiographs have been obtained, or these can be collected prospectively in window per schedule of events
   * 12-month post-operative KOOS JR have been obtained, or these can be collected prospectively in window per schedule of events
2. Subject's treating clinician has decided the study device is suitable for the subjects TKA procedure and the study device is used in line with the applicable Instructions For Use (IFU) (listed in section 6).
3. Subject agrees to consent and follow the prospective study visit schedule up to 10 years post-surgery (as defined in the study protocol and informed consent form) by signing the Independent Review Board (IRB)/Independent Ethics Committee (IEC) approved consent form.
4. Subject is able to read, understand and communicate responses to Patient Reported Outcome Measure (PROM).
5. Subject is 18-80 years old at the time of consent (inclusive).

Exclusion Criteria:

1. Subject received revision TKA on the contralateral knee for a previously failed TKA, or Unicondylar Knee Arthroplasty (UKA).
2. Subject has a Body Mass Index (BMI) ≥ 40 at pre-operative visit.
3. Subject has ipsilateral hip arthritis resulting in flexion contracture of the hip joint.
4. At the time of surgery, subject has one or more of the following arthroplasties that are not fully healed and/or well-functioning, in the opinion of the Investigator: Ipsilateral or contralateral primary total hip arthroplasty or hip resurfacing arthroplasty; contralateral primary TKA or UKA.
5. Subject has a condition that may interfere with the TKA survival or outcome (e.g., Paget's or Charcot's disease, vascular insufficiency, lupus, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease).
6. Subject has a known allergy to one or more of the components of the study device.
7. Any subject with hardware present in ipsilateral distal femur or proximal tibia.
8. Any subject that meets the definition of a Vulnerable Subject per ISO 14155 Section 3.55.
9. Subject is entered in another drug, biologic, or device study or has been treated with an investigational product in the past 30 days (30 days from operation/dosing).
10. Subject, in the opinion of the Investigator, has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study, ability to consent or complete the PROMs, including mental illness, drug or alcohol abuse.
11. In the opinion of the Investigator, or site staff, Subject is at risk for lost to follow-up, or failure to return for scheduled visits.
12. Women who are pregnant, nursing, or of child-bearing potential who are not utilizing highly effective birth control measures at the time of screening or the time of surgery.
13. Subjects who have participated previously in this clinical trial and who have been withdrawn.
14. Subject does not meet the indication or is contraindicated for TKA according to specific Smith+Nephew LEGION Knee System IFU.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants needing primary Total Knee Arthroplasty (TKA) due to degenerative joint disease (primary diagnosis of osteoarthritis), post-traumatic arthritis or inflammatory arthritis.
  OR
  Participants which have undergone primary TKA using the investigational product in the past 12 months to repair degenerative joint disease, post-traumatic arthritis or inflammatory arthritis and all the following conditions have been met:
  * Pre-operative Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS JR) has been obtained
  * Post-operative radiographs have been obtained, or these can be collected prospectively in window per schedule of events
  * 12-month post-operative KOOS JR have been obtained, or these can be collected prospectively in window per schedule of events
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2036-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
Implant Survivorship at 10 Years | 10 years
  Implant survivorship at 10 years post-surgery. Implant survivorship is defined as the cumulative proportion of knee-implanted components without a revision. Survivorship is defined as absence of revision of any, or all, of the tibial / femoral / insert components that were implanted during the primary TKA - not including the patella.
  (Revision is the removal of some, or all, of the above specified implant components, and replacement with new ones for any reason).

SECONDARY OUTCOMES:
Implant Survivorship | 6 weeks, 1 year, 2 years, 3 years, 5 years, and 7 years
  Implant survivorship at 6 weeks, 1, 2, 3, 5, 7 years post-surgery. Implant survivorship is defined as the cumulative proportion of knee-implanted components without a revision. Survivorship is defined as absence of revision of any, or all, of the tibial / femoral / insert components that were implanted during the primary TKA - not including the patella.
  (Revision is the removal of some, or all, of the above specified implant components, and replacement with new ones for any reason).
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS JR) | 6 weeks, 1 year, 2 years, 3 years, 5 years, 7 years, and 10 years
  The Knee injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR) is a validated short form of the KOOS that assesses patient stiffness (1 item), pain (4 items), and functions of daily living (2 items). Scores range from 0 to 100 with a score of 0 indicating total knee disability (i.e., worse outcome) and 100 indicating perfect knee health (i.e., better outcome).
Oxford Knee Score (OKS) | 6 weeks, 1 year, 2 years, 3 years, 5 years, 7 years, and 10 years
  The OKS consists of twelve questions covering function and pain associated with the knee. Scores from the twelve questions are combined to provide an overall score that ranges from 0 to 48, with higher scores indicating better knee function and less pain (i.e., a better outcome)
Forgotten Joint Score (FJS) | 6 weeks, 1 year, 2 years, 3 years, 5 years, 7 years, and 10 years
  The Forgotten Joint Score (FJS) is a patient reported outcome that focuses on the participant's awareness of a specific joint in everyday life. Joint awareness can be simply defined as any unintended perception of a joint. Scores are on a scale of 1 to 100, with higher scores indicating a better outcome.
Five-Level EuroQol Five-Dimensional (EQ-5D-5L): Index Score | 6 weeks, 1 year, 2 years, 3 years, 5 years, 7 years, and 10 years
  The EQ-5D-5L score consists of two parts: a descriptive system and a visual analogue scale (VAS). The descriptive system (i.e., index score) is used to describe the participant's health state and consists of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels to choose the most appropriate answer: no problems, slight problems, moderate problems, severe problems and extreme problems. The participant is asked to indicate their health state by marking the most appropriate statement in each of the five areas. The EQ-5D-5L Index Score was based on a scale of 0 to 1, with higher index values indicating better health and lower index values indicating worse health.
Five-Level EuroQol Five-Dimensional (EQ-5D-5L): Visual Analogue Scale Score | 6 weeks, 1 year, 2 years, 3 years, 5 years, 7 years, and 10 years
  The EQ-5D-5L score consists of two parts: a descriptive system and a visual analogue scale (VAS). The VAS records the participant's self-rated health on a vertical visual analogue scale. The scale ranges from 0 to 100 where 0 indicates 'The worst health you can imagine' and 100 indicates 'The best health you can imagine'.

CONTACTS AND LOCATIONS:
Overall Officials: Anasua Ganguly, Study Chair — Smith & Nephew, Inc.
Locations (6):
- United States (6):
  - The Core Institute, Phoenix, Arizona
  - Rothman Orthopedics-Advent Health, Orlando, Florida
  - Newton Wellesley Hospital, Newton, Massachusetts
  - New York University Hospital, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No